CLINICAL TRIAL: NCT01995253
Title: A Smartphone Application to Evaluate Energy Expenditure and Duration of Moderate-intensity Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Almerys (Other)
Responsible Party: Principal Investigator, Martine DUCLOS, PUPH, University Hospital, Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AU979; 2012-A00809-34 (Other: ANSM)
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2013-11

CONDITIONS: Accelerometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Controlled conditions (Experimental)
  Interventions: Device: Energy expenditure estimation in controlled conditions
- Free-living conditions (Experimental)
  Interventions: Device: Energy expenditure estimation in free-living conditions

INTERVENTIONS:
Device: Energy expenditure estimation in controlled conditions — Volunteers were asked to perform several activities such as walking at different paces, running, sitting, standing still or taking public transportation for about 3h30 They wore 2 research sensors that estimate energy expenditure: Armband and Actiheart. They also wore a smartphone (in a front pant pocket) that collected accelerometry data.
  Arms: Controlled conditions
Device: Energy expenditure estimation in free-living conditions — Volunteers were asked to wear sensors during about 12 hours, one day. They wore 2 research sensors that estimate energy expenditure: Armband and Actiheart. They also wore a smartphone (in a front pant pocket) that collected accelerometry data.
  Arms: Free-living conditions

SUMMARY:
The aim of this study was to find functions for estimating energy expenditure in free-living conditions. This method was based on accelerometry data acquired from a smartphone worn in a trouser pocket. The developed functions have been compared to the estimations provided by two research devices named Armband and Actiheart.

DETAILED DESCRIPTION:
There is a growing interest in evaluating physical activity and energy expenditure (EE) to provide feedback to the user. The use of mass-market sensors such as accelerometers offers a promising solution for the general public due to the growing smartphone market over the last decade.

Thus, the proposed EE estimation function has been created using accelerometry data collected from 10 volunteers equipped with a smartphone and two research sensors (Armband and Actiheart) used to estimate EE during several controlled activities. The research sensors' data serves as reference during the creation and evaluation of the proposed function.

It has been evaluated with data of 6 other volunteers in free-living conditions. This new EE function using the smartphone technology is dedicated to light- and moderate-intensity activities, and we believe it can be a new way to help people controlling their daily physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* age: 18-60 years
* BMI between 18.5 and 25 kg/m²
* subject considered as healthy after clinical examination and medical questionnaire
* women of childbearing age: negative beta-HCG
* subject with normal rest electrocardiogram (validated by a cardiologist)
* subject with normal blood pressure (<140/90 mm Hg) with or without medical treatment
* subject with no foot pad problem
* subject giving his/her written informed consent
* subject willing to comply with study procedures
* affiliated to National Health Insurance

Exclusion Criteria:

* respiratory failure or cardiovascular problem
* known cardiac decompensation or myocardial infarction
* surgery made less than 6 months before the study beginning
* pregnant women and nursing mother
* current infectious pathology
* abnormal electrocardiogram
* not affiliated to national health insurance people
* under legal guardianship
* refusal to sign informed consent
* refusal to be registered on the national volunteers data file
* currently participating or who having got 4500€ in this year before to have participated in another clinical trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Accelerometry | about 17Hz (duration: 3h30 in controlled conditions; 12 hours in free-living conditions)
  Measures acquired by a smartphone (it contains several sensors, including a tri-axial accelerometer)

SECONDARY OUTCOMES:
Energy expenditure | one point recorded each minute for 3h30 in controlled conditions or 12 hours in free-living conditions
  Sensor: Armband
Energy expenditure | one point recorded each minute for 3h30 in controlled conditions or 12 hours in free-living conditions
  Sensor: Actiheart

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche en Nutrition Humaine Auvergne, Clermont-Ferrand, France